CLINICAL TRIAL: NCT06307626
Title: A Phase 3, Randomized, Double-Masked, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Efgartigimod PH20 SC Administered by Prefilled Syringe in Adult Participants With Thyroid Eye Disease
Brief Title: A Study of Efgartigimod PH20 SC Given by Prefilled Syringe in Adults With Thyroid Eye Disease.
Acronym: UplighTED
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2309; 2023-509198-22-00 (EU CTIS Number)
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod arm (Experimental): Participants with active, moderate-to-severe TED receiving Efgartigimod PH20 SC (subcutaneously) via pre-filled syringe (PFS)
  Interventions: Combination Product: Efgartigimod PH20 SC
- Placebo arm (Placebo Comparator): Participants with active, moderate-to-severe TED receiving Placebo PH20 SC (subcutaneously) via pre-filled syringe (PFS)
  Interventions: Other: Placebo PH20 SC

INTERVENTIONS:
Combination Product: Efgartigimod PH20 SC — Subcutaneous efgartigimod PH20 SC given by prefilled syringe
  Arms: Efgartigimod arm
Other: Placebo PH20 SC — Subcutaneous placebo given by prefilled syringe
  Arms: Placebo arm

SUMMARY:
This study aims to evaluate the efficacy, safety and tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and immunogenicity of efgartigimod PH20 SC in participants with active, moderate-to-severe TED, compared with placebo PH20 SC.

After the screening period, eligible participants will be randomized in a 2:1 ratio to receive efgartigimod PH20 SC or placebo PH20 SC, respectively during the double-blinded treatment period (DBTP). At the end of the DBTP, participants may enter a follow-up observational period while off study drug. Some participants may also enter the open-label treatment period with efgartigimod PH20 SC. The study duration varies from approximately 60 to 110 weeks.

An alternative list of clinical sites open for recruitment could be found in the other UplighTED study record (https://www.clinicaltrials.gov/study/NCT06307613).

This study was terminated early on 15 December 2025 as the pre-defined interim analysis concluded that continuing the trials is unlikely to demonstrate the intended efficacy. This decision is not related to safety concerns, and the safety profile of efgartigimod remains unchanged. End-of-study and Safety-Follow-Up visits are ongoing for the participants of this trial.

ELIGIBILITY:
Inclusion Criteria:

* The participant is at least 18 years of age
* The participant is capable of providing signed informed consent and following with protocol requirements
* The investigator determines active, moderate-to-severe thyroid eye disease (TED) associated with autoimmune thyroid conditions (Graves' disease or Hashimoto's thyroiditis) for the most severely affected eye
* The participant has first onset of active TED symptoms within 12 months before screening
* The participant must have normal thyroid function with the baseline disease under control or have mild hypo or hyperthyroidism at screening. Every effort should be made to correct the mild hypo or hyperthyroidism promptly and to maintain the normal thyroid function for the full duration of the study
* The participant agrees to use birth control consistent with local regulations and the people of child-bearing potential must have a negative blood pregnancy test at screening and a negative urine pregnancy test before receiving the study drug

Exclusion Criteria:

* Optic neuropathy (damage to optic nerve), defined as new visual field defect (blind spot), relative afferent pupillary defect (pupils respond differently to light), or color defect secondary to optic nerve involvement within the 6 months before screening
* Corneal decompensation (swelling of the cornea) unresponsive to medical management
* Previous orbital irradiation or surgery for TED
* Use of some medications before screening (more information is found in the protocol)
* Known autoimmune disease or any medical condition that would interfere with an accurate assessment of clinical symptoms of TED or puts the participant at undue risk
* History of malignancy, cancer, unless considered cured by adequate treatment with no evidence of recurrence for ≥3 years. Adequately treated participants with the following cancers can be included at any time: Basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histological findings of prostate cancer
* Clinically significant active infection that is not sufficiently resolved in the investigator's opinion or positive serum test at screening for active infection with any of the following: Hepatitis B virus (HBV), Hepatitis C virus (HCV), HIV
* Current participation in another interventional clinical study or previous participation in an efgartigimod clinical study and at least 1 dose of study drug received or has received at least 1 dose of commercially available efgartigimod
* Known hypersensitivity to study drug or one of its excipients (inactive ingredients)
* History of or current alcohol, drug, or medication abuse within 12 months before screening as assessed by the investigator
* Pregnant or lactating state or intention to become pregnant during the study
* Live or live-attenuated vaccine received <4 weeks before screening

The complete list of exclusion criteria can be found in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who were proptosis responders | At week 24 of the Double-Blinded Treatment Period

SECONDARY OUTCOMES:
Change in proptosis measurement in the study eye from baseline | Up to week 24 of the Double-Blinded Treatment Period
Change in the total Graves' Orbitopathy Quality of Life (GO-QoL) score from baseline | Up to week 24 of the Double-Blinded Treatment Period
  Minimum value: 0 (most negative impact on Quality of Life); Maximum value: 100 (No impact on Quality of Life)
Percentage of participants with a resolution of diplopia (responders) | At week 24 of the Double-Blinded Treatment Period

CONTACTS AND LOCATIONS:
Locations (76):
- United States (11):
  - American Institute of Research, Los Angeles, California
  - North Valley Eye Medical Group, Inc., Mission Hills, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Cockerham Eye Consultants, San Diego, California
  - Sibia Eye Institute, Boynton Beach, Florida
  - Sarasota Retina Institute (SRI), Sarasota, Florida
  - Butchertown Clinical Trials, Louisville, Kentucky
  - St. Louis University (SLU) Care - Center for Specialized Medicine, St Louis, Missouri
  - Advancing Research International, LLC, Las Vegas, Nevada
  - New York Eye & Ear Infirmary, New York, New York
  - Baylor College of Medicine, Houston, Texas
- Austria (2):
  - Landeskrankenhaus - Universitaetskliniken Innsbruck, Innsbruck
  - Hanusch-Krankenhaus - Vienna Institute for Research in Ocular Surgery, Vienna
- Bulgaria (4):
  - AIPSMAED Sveti Luka EOOD, Plovdiv
  - Multi-Profile Hospital for Active Treatment (MHAT) Hadji Dimitar, Sliven
  - Medical Center Hera EOOD, Sofia
  - Military Medical Academy (MMA), Sofia
- China (6):
  - Peking University Third Hospital, Beijing
  - The Second Affiliated Hospital of Chengdu Medical College / Nuclear Industry 416 Hospital, Chengdu
  - The Second Hospital of Dalian Medical University, Dalian
  - Fujian Provincial Hospital, Fuzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Shandong Provincial Hospital of Shandong First Medical University, Jinan
- France (4):
  - Hospices Civils de Lyon (HCL) - Hopital Louis Pradel, Bron
  - CHU Lille - Hopital Huriez, Lille
  - Centre Hospitalier National d'Ophtalmologie (Chno) Des Quinze-Vingts, Paris
  - CHU de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
- Georgia (4):
  - JSC Curatio, Tbilisi
  - National Institute of Endocrinology, Tbilisi
  - New Hospitals, Tbilisi
  - Caucasus Medical Centre, Tbilisi
- Germany (4):
  - Universitaetsklinikum Essen (AoR), Essen
  - Klinikum Der Albert-Ludwigs Universitaet Freiburg, Freiburg im Breisgau
  - Philipps-Universitaet Marburg Universitaetsklinikum Giessen und Marburg Klinik fuer Augenheilkunde, Marburg
  - Universitaetsaugenklinik Ulm, Ulm
- Italy (5):
  - Universita degli Studi di Cagliari - Ospedale San Giovanni di Dio, Cagliari
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele (HSR) (Istituto Scientifico Universitario San Raffaele), Milan
  - Ospedale Cisanello, Pisa
  - Azienda Ospedaliero Universitaria Sant'Andrea, Roma
  - Azienda Ospedaliero Ordine Mauriziano Torino - Ospedale Umberto I di Torino, Torino
- Japan (12):
  - Kanazawa University Hospital, Kanazawa
  - Hospital of University of Occupational and Environmental Health, Kitakyushu
  - Shinkoga clinic, Kurume
  - Koga Hospital Group - Shinkoga Hospital, Kurume-shi
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Kozawa Eye Hospital and Diabetes Center, Mito
  - Nagasaki University Hospital, Nagasaki
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka City General Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - Tohoku Medical and Pharmaceutical University - Fukumuro, Sendai
  - Tottori University Hospital, Yonago
- Latvia (2):
  - Daugavpils Regionala Slimnica, Daugavpils
  - Paula Stradina Kliniska universitates slimnica, Riga
- Poland (6):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Centrum Medycyny Inwazyjnej, Gdansk
  - Szpital Sw. Rozy, Krakow
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Centrum Zdrowia MDM, Warsaw
- Clinical Center Vojvodina, Novi Sad, Serbia
- Slovenia (2):
  - OLHB d.o.o., Ljubljana
  - University Medical Centre University Eye Hospital, Ljubljana
- Spain (4):
  - Institut Catala de Retina (ICR) Centre Oftalmologic - ICR Seu Central Ganduxer, Barcelona
  - Hospital La Arruzafa, Córdoba
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Eye Clinic Linkoping, Linköping, Sweden
- Switzerland (2):
  - Universitaetsspital Bern - Inselspital, Bern
  - ADMEDICO Augenzentrum AG, Olten
- Turkey (Türkiye) (2):
  - Memorial Ankara Hospital, Ankara
  - Kocaeli University Research and Training Hospital, Kocaeli
- United Kingdom (4):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Royal Liverpool University Hospital , St Paul's Eye Unit - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Moorfields Eye Hospital, London
  - Western Eye Hospital - Imperial College Healthcare NHS Trust, London